CLINICAL TRIAL: NCT06358404
Title: Developing a Peer Support Intervention for Depression in SCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jin hui Joo, MD, MA, Assistant Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024P000615
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2025-05-12 (Actual); Status verified 2025-05

CONDITIONS: Subjective Cognitive Decline; Depression in Old Age

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Peer coaches will deliver the PeersCOG intervention to participants.
  Interventions: Behavioral: PeersCOG

INTERVENTIONS:
Behavioral: PeersCOG — . The intervention will consist of 8 weekly video chats focused on emotional, appraisal, and informational support delivered by community-based older adult peer coaches to adults 60 years of age and older with subthreshold depression and SCD.

SUMMARY:
The purpose of this study is to assess the feasibility, acceptability, and fidelity of an 8-week intervention where peer coaches will deliver depression care to adults 60 years of age or older who have depression and subjective cognitive decline.

DETAILED DESCRIPTION:
With support from the MADRC ORE Core, we will recruit 30 community-dwelling older adults to conduct an open pilot study of PeersCOG. Trained and supervised peer coaches will deliver depression care to adults 60 years of age and older with depression and subjective cognitive decline in an 8-week intervention using video chats and texts. We will use mixed methods to assess feasibility, acceptability, and fidelity. We will use validated instruments to assess the preliminary outcomes, including depression, SCD, functioning, and social factors at baseline, 8 weeks, and 3 months, and we will conduct post-intervention interviews with stakeholders at 8 weeks. Older adult participants will be asked to name a study partner who will support the older adult throughout the study in terms of study enrollment. They may also have additional perspectives on the impact of impaired cognition and depression on daily living and related needs. The older adult will not be excluded if the study partner is not available.

ELIGIBILITY:
Inclusion Criteria:

* Older adults aged 60+
* Endorse subjective cognitive decline
* Endorse depressive symptoms
* not currently experiencing suicidal ideation nor active, untreated manic, psychotic, or substance use disorder
* fluent in English and able to give informed consent

Exclusion Criteria:

* Meets diagnostic criteria for mild cognitive impairment or Alzheimer's dementia
* Meets diagnostic criteria for a current major depressive disorder
* have a history of neurological and psychiatric comorbidities such as major depressive disorder in the past 12 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention | Measured at baseline enrollment
  Level of participant engagement: how many screened older adults agree to participate in the intervention and complete baseline assessments
Acceptability of Intervention | Measured during intervention (8 weeks)
  Number of meetings older adults complete with peer coach
Fidelity of Intervention | Measured during intervention (8 weeks)
  Degree of adherence to intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States